CLINICAL TRIAL: NCT03314662
Title: A Phase 3, Randomized, Double-Blind, Controlled, Multicenter, Clinical Study to Evaluate Safety and Immunogenicity of an MF59-Adjuvanted Quadrivalent Subunit Influenza Vaccine in Comparison With an MF59-Adjuvanted Trivalent Subunit Influenza Vaccine and an MF59-Adjuvanted Trivalent Subunit Influenza Vaccine Containing the Alternate B Strain, in Adults Aged 65 Years and Above
Brief Title: Phase 3 Safety and Immunogenicity Study of aQIV in Elderly Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V118_20
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial is designed as a double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- aQIV (Experimental): MF59-adjuvanted Quadrivalent Subunit Inactivated Egg-derived Influenza Vaccine (aQIV) contains each of the 2 influenza type A strains and each of the two influenza type B strains in the vaccine.
  Interventions: Biological: MF59-adjuvanted Quadrivalent Subunit Inactivated Egg-derived Influenza Vaccine (aQIV)
- aTIV-1 (Experimental): Licensed MF59-adjuvanted Trivalent Subunit Inactivated Egg-derived Influenza Vaccine (aTIV-1) contains each of the 2 influenza type A strains and one influenza type B strain in the vaccine.
  Interventions: Biological: Licensed MF59-adjuvanted Trivalent Subunit Inactivated Egg-derived Influenza Vaccine (aTIV-1)
- aTIV-2 (Experimental): MF59-adjuvanted Trivalent Subunit Inactivated Egg-derived Influenza Vaccine contains each of the 2 influenza type A strains and alternate influenza type B strain in the vaccine.
  Interventions: Biological: MF59-adjuvanted Trivalent Subunit Inactivated Egg-derived Influenza Vaccine Containing the Alternate B Strain (aTIV-2)

INTERVENTIONS:
Biological: MF59-adjuvanted Quadrivalent Subunit Inactivated Egg-derived Influenza Vaccine (aQIV) — The strain composition is that recommended by the World Health Organization for the 2017-2018 Northern Hemisphere influenza season (WHO, 2017) for quadrivalent vaccines.
  Arms: aQIV
Biological: Licensed MF59-adjuvanted Trivalent Subunit Inactivated Egg-derived Influenza Vaccine (aTIV-1) — The strain composition is that recommended by the World Health Organization for the 2017-2018 Northern Hemisphere influenza season (WHO, 2017) for trivalent vaccines.
  Arms: aTIV-1
Biological: MF59-adjuvanted Trivalent Subunit Inactivated Egg-derived Influenza Vaccine Containing the Alternate B Strain (aTIV-2) — The strain composition is that recommended by the World Health Organization for the 2017-2018 Northern Hemisphere influenza season (WHO, 2017) for trivalent vaccines except the B strain present in this vaccine is the second/alternate B strain recommended for inclusion in quadrivalent vaccines (ie, Alternate B strain).
  Arms: aTIV-2

SUMMARY:
This phase 3 study is a randomized, double-blinded, comparator controlled, parallel-group, multicenter study of aQIV versus the US-licensed 2017-2018 adjuvanted trivalent influenza vaccine (aTIV-1, Fluad), and versus an adjuvanted trivalent influenza vaccine (aTIV-2), containing the alternate B strain.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 65 years old who are healthy or have co-morbidities
* Individuals who or whose legal representative(s) have voluntarily given written consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry
* Ability to attend all scheduled visits and to comply with study procedures including diary card completion and follow-up

Exclusion Criteria:

* History of behavioral or cognitive impairment or psychiatric condition
* Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study
* Abnormal function of the immune system
* Receipt of any influenza vaccine within 6 months prior to enrollment in this study, or plan to receive influenza vaccine prior to the Day 22 blood collection
* Any other clinical condition that, in the opinion of the Investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study

Additional eligibility criteria may be discussed by contacting the site.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1778 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Scientist, Study Director — Seqirus
Locations (20):
- United States (20):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Anaheim Clinical Trials, Anaheim, California
  - Paradigm clinical Research Centers, Inc, Redding, California
  - Clinical Research of South Florida, an AMR Company, Coral Gables, Florida
  - Meridan Clinical Research, LLC, Savannah, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Heartland Research Associates, LLC - An AMR Company, Newton, Kansas
  - Heartland Research Associates, LLC - An AMR Company, Wichita, Kansas
  - Center for Pharmaceutical Research, LLC, Kansas City, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - United Medical Associates, Binghamton, New York
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Medical Research South, Charleston, South Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Benchmark Research, Fort Worth, Texas
  - Benchmark Research, San Angelo, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Essink B, Fierro C, Rosen J, Figueroa AL, Zhang B, Verhoeven C, Edelman J, Smolenov I. Immunogenicity and safety of MF59-adjuvanted quadrivalent influenza vaccine versus standard and alternate B strain MF59-adjuvanted trivalent influenza vaccines in older adults. Vaccine. 2020 Jan 10;38(2):242-250. doi: 10.1016/j.vaccine.2019.10.021. Epub 2019 Oct 18. PMID 31635976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 study centers in the United States
Pre-assignment Details: All enrolled subjects were randomized.
Groups:
- aQIV: MF59-adjuvanted Quadrivalent Subunit Inactivated Egg-derived Influenza Vaccine (aQIV) contains each of the 2 influenza type A strains and each of the two influenza type B strains in the vaccine.The strain composition is that recommended by the World Health Organization for the 2017-2018 Northern Hemisphere influenza season (WHO, 2017) for quadrivalent vaccines.
- aTIV-1: Licensed MF59-adjuvanted Trivalent Subunit Inactivated Egg-derived Influenza Vaccine (aTIV-1) contains each of the 2 influenza type A strains and one influenza type B strain in the vaccine.The strain composition is that recommended by the World Health Organization for the 2017-2018 Northern Hemisphere influenza season (WHO, 2017) for trivalent vaccines.
- aTIV-2: MF59-adjuvanted Trivalent Subunit Inactivated Egg-derived Influenza Vaccine contains each of the 2 influenza type A strains and alternate influenza type B strain in the vaccine.The strain composition is that recommended by the World Health Organization for the 2017-2018 Northern Hemisphere influenza season (WHO, 2017) for trivalent vaccines except the B strain present in this vaccine is the second/alternate B strain recommended for inclusion in quadrivalent vaccines (ie, Alternate B strain).
Period: Overall Study
Arm/Group | aQIV | aTIV-1 | aTIV-2
Started | 889 | 445 | 444
Treated | 888 | 444 | 444
Completed | 881 | 440 | 439
Not Completed | 8 | 5 | 5
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Lost to Follow-up | 5 | 4 | 4
Not completed — Death | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- aQIV: MF59-adjuvanted Quadrivalent Subunit Inactivated Egg-derived Influenza Vaccine (aQIV) contains each of the 2 influenza type A strains and each of the two influenza type B strains in the vaccine. The strain composition is that recommended by the World Health Organization for the 2017-2018 Northern Hemisphere influenza season (WHO, 2017) for quadrivalent vaccines.
- aTIV-1: Licensed MF59-adjuvanted Trivalent Subunit Inactivated Egg-derived Influenza Vaccine (aTIV-1) contains each of the 2 influenza type A strains and one influenza type B strain in the vaccine. The strain composition is that recommended by the World Health Organization for the 2017-2018 Northern Hemisphere influenza season (WHO, 2017) for trivalent vaccines.
- Total: Total of all reporting groups
Arm/Group | aQIV | aTIV-1 | aTIV-2 | Total
Number analyzed (Participants) | 889 | 445 | 444 | 1778
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (5.54) | 72.4 (5.60) | 72.6 (5.46) | 72.5 (5.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 517 | 249 | 241 | 1007
  Male | 372 | 196 | 203 | 771
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 814 | 403 | 411 | 1628
  Black or African American | 59 | 37 | 29 | 125
  Asian | 9 | 2 | 1 | 12
  Native Hawaiian or Pacific Islander | 1 | 1 | 0 | 2
  American Indian or Alaska Native | 5 | 0 | 2 | 7
  Other | 1 | 2 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 37 | 31 | 127
  Not Hispanic or Latino | 827 | 408 | 410 | 1645
  Not Reported | 2 | 0 | 2 | 4
  Unknown | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 889 | 445 | 444 | 1778
Height [Mean (Standard Deviation); unit: cm] — Population: analysis presented for subjects with available data.
  cm
    number analyzed (Participants) | 885 | 442 | 444 | 1771
    (all) | 167.54 (9.350) | 167.92 (10.535) | 168.38 (10.646) | 167.84 (9.990)
Weight [Mean (Standard Deviation); unit: kg] — Population: analysis presented for subjects with available data.
  kg
    number analyzed (Participants) | 885 | 442 | 444 | 1771
    (all) | 83.24 (19.064) | 84.18 (8.963) | 84.24 (17.825) | 83.73 (18.731)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: analysis presented for subjects with available data.
  kg/m^2
    number analyzed (Participants) | 885 | 442 | 444 | 1771
    (all) | 29.60 (6.157) | 29.79 (5.858) | 29.69 (5.647) | 29.67 (5.956)
Influenza Vaccination History [Count of Participants; unit: Participants]
  No | 129 | 65 | 43 | 237
  Yes | 760 | 380 | 401 | 1541
Total Risk Score (Comorbidity) [Mean (Standard Deviation); unit: units on a scale] — Comorbidity risk scores were assessed among other baseline characteristics and validated the risk of influenza complications in subjects ≥65 y.o. This model-based approach assessed 5 classifications: pulmonary disease, heart disease, renal disease, dementia or stroke, and non-hematological and hematological cancer [excl. cancer of the skin other than melanoma]).
  The score(s) include: <50 (low risk) to ≥50 (high risk for hospitalization due to pneumonia or influenza and death from any cause).
  The outer ranges of the comorbidity scale (i.e., min and max) are below:
  0 (min.) to 267 (max.)
  units on a scale | 46.0 (33.50) | 44.6 (30.25) | 46.5 (34.15) | 45.8 (32.88)

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity Endpoint: The Geometric Mean Titer (GMT) and GMT Ratio for the Four Strains Included in the Vaccine, Non-inferiority Analysis.
Description: The GMT of the post-vaccination (Day 22) hemagglutination inhibition (HI) titer. The GMT ratio was defined as the GMT for aTIV-1 (or aTIV-2) over the GMT for aQIV for all of the four strains.
Time Frame: Day 22
Population: The per protocol set (PPS) Immunogenicity comprised all subjects who were randomized, received at least 1 study vaccination, and provided immunogenicity data at Day 1 and Day 22, and who did not have any major protocol deviations that were assessed as potentially impacting on immunogenicity results
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titer
Groups:
- aQIV: MF59-adjuvanted Quadrivalent Subunit Inactivated Egg-derived Influenza Vaccine (aQIV) contains each of the 2 influenza type A strains and each of the 2 influenza type B strains in the vaccine. The strain composition is that recommended by the World Health Organization for the 2017-2018 Northern Hemisphere influenza season (WHO, 2017) for quadrivalent vaccines.
- aTIV-2: MF59-adjuvanted Trivalent Subunit Inactivated Egg-derived Influenza Vaccine (aTIV-2) contains each of the 2 influenza type A strains and alternate influenza type B strain in the vaccine. The strain composition is that recommended by the World Health Organization for the 2017-2018 Northern Hemisphere influenza season (WHO, 2017) for trivalent vaccines except the B strain present in this vaccine is the second/alternate B strain recommended for inclusion in quadrivalent vaccines (ie, Alternate B strain).
- aTIV-1/aTIV-2: Pooled Subjects Treated with aTIV-1 and aTIV-2
Arm/Group | aQIV | aTIV-1 | aTIV-2 | aTIV-1/aTIV-2
Number analyzed (Participants) | 872 | 436 | 433 | 869
Geometric mean titer
  A/H1N1 | 65.01 [57.79 to 73.13] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 75.16 [66.68 to 84.72]
  A/H3N2 | 294.91 [261.88 to 332.09] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 293.31 [259.91 to 330.99]
  B/Yamagata | 24.67 [22.67 to 26.84] | 15.96 [14.48 to 17.59] | 24.30 [22.00 to 26.84] | NA [NA to NA] — Analysis was not performed
  B/Victoria | 30.78 [28.27 to 33.51] | 30.13 [27.31 to 33.24] | 21.80 [19.73 to 24.09] | NA [NA to NA] — Analysis was not performed
Statistical Analysis 1: Comparison: aQIV vs aTIV-1 vs aTIV-2; Comparison Group Selection: aTIV/aQIV - for strain A/H1N1; Test type: Non-Inferiority — aQIV was considered non-inferior to aTIV-1 or aTIV-2 if the upper bound of the two-sided 95% confidence interval (CI) for the ratios of GMTs (aTIV/aQIV) do not exceed 1.5; GMT ratio (aTIV/aQIV) = 1.16, 95% CI 2-sided [1.05 to 1.27] — GMT ratios (adjusted) obtained from a GLM fitted on log-transformed (base 10) post-vaccination HI titer as outcome variable and covariate terms: treatment, pre-vaccination HI titer (log10 transformed), age, sex, vaccination history, study site
Statistical Analysis 2: Comparison: aQIV vs aTIV-1 vs aTIV-2; Comparison Group Selection: aTIV/aQIV - performed for strain A/H3N2; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMT ratio: (aTIV/aQIV = 0.99, 95% CI 2-sided [0.90 to 1.09] — GMT ratios (adjusted) obtained from a GLM fitted on log-transformed (base 10) post-vaccination HI titer as outcome variable and covariate terms: treatment, pre-vaccination HI titer (log 10 transformed), age, sex, vaccination history, study site
Statistical Analysis 3: Comparison: aQIV vs aTIV-1 vs aTIV-2; Comparison Group Selection: aQIV/aTIV - performed for strain B/Yamagata; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMT ratio: aTIV/aQIV = 0.99, 95% CI 2-sided [0.90 to 1.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: aQIV vs aTIV-1 vs aTIV-2; Comparison Group Selection: aQIV/aTIV - performed for strain B/Victoria; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMT ratio: (aTIV/aQIV)] = 0.98, 95% CI 2-sided [0.89 to 1.08] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Immunogenicity Endpoint: The Difference Between the Seroconversion Rate (SCR) for the Four Strains Included in the Vaccine, Non-inferiority Analysis
Description: The SCR is defined as the percentage of subjects with either a pre-vaccination HI titer < 1:10 and a post-vaccination HI titer >= 1:40 or a pre-vaccination HI titer >= 1:10 and a >= 4-fold increase in post-vaccination HI titer. The SCR Difference is defined as the difference between the SCR of post- vaccination (Day 22) HI titer for aTIV-1 (or aTIV-2) and the SCR of post-vaccination (Day 22) HI titer for aQIV. aTIV-1 and aTIV-2 vaccine groups are pooled for the analysis of A-H1N1 and A-H3N2 strains. For B/Victoria TIV=TIV-1. For B/Yamagata TIV=TIV-2.
Time Frame: Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV | aTIV-1 | aTIV-2
Number analyzed (Participants) | 872 | 436 | 433
percentage of subjects
  A/H1N1 | 35.21 [32 to 38.5] | 39.45 [34.8 to 44.2] | 37.41 [32.8 to 44.2]
  A/H3N2 | 39.33 [36.1 to 42.7] | 39.70 [36.4 to 43.0] | 37.18 [32.6 to 41.9]
  B/Yamagata | 16.4 [14.0 to 19.0] | NA [NA to NA] — Not applicable as the strain is not present in aTIV vaccine | 15.47 [12.2 to 19.2]
  B/Victoria | 13.42 [11.2 to 15.9] | 12.16 [9.24 to 15.6] | NA [NA to NA] — Not applicable as the strain is not present in aTIV vaccine
Statistical Analysis 1: Comparison: aQIV vs aTIV-1 vs aTIV-2; Comparison Group Selection: aTIV minus aQIV - for strain A/H1N1; Test type: Non-Inferiority — aQIV was considered non-inferior to aTIV-1 or aTIV-2 if the upper bound of the two-sided 95% CI for the differences between the SCRs (aTIV - aQIV) do not exceed 10% for each of the four strains; SCR difference (aTIV minus aQIV) = 3.23, 95% CI 2-sided [-1.30 to 7.76]
Statistical Analysis 2: Comparison: aQIV vs aTIV-1 vs aTIV-2; Comparison Group Selection: aTIV minus aQIV - for strain A/H3N2; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; SCR difference (aTIV minus aQIV) = 0.37, 95% CI 2-sided [-4.23 to 4.96]
Statistical Analysis 3: Comparison: aQIV vs aTIV-1 vs aTIV-2; Comparison Group Selection: aTIV minus aQIV - for strain B-Yamagata; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; SCR difference (aTIV minus aQIV)] = -0.93, 95% CI 2-sided [-5.13 to 3.27]
Statistical Analysis 4: Comparison: aQIV vs aTIV-1 vs aTIV-2; Comparison Group Selection: aTIV minus aQIV - for strain B-Victoria; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Other [SCR difference (aTIV minus aQIV)] = -1.26, 95% CI 2-sided [-5.07 to 2.55]

3. Primary Outcome: Immunogenicity Endpoint: The Percentage of Subjects Achieving SCR for Hemagglutination Inhibition (HI) Antibody for the Four Strains Included in the Vaccine.
Description: The percentage of subjects vaccinated with aQIV achieving SCR at Day 22 was assessed for each of the 4 strains. SCR was defined as the percentage of subjects with either a pre-vaccination HI titer <1:10 and a post-vaccination HI titer ≥1:40 or a pre-vaccination HI titer ≥1:10 and a ≥4-fold increase in post-vaccination HI titer. Assessment criteria was considered fulfilled if the lower bound of the two-sided 95% confidence interval for the percentage of subjects achieving SCR for HI antibody should meet or exceed 30%.
Time Frame: Day 22
Population: The PPS Immunogenicity comprised all subjects who were randomized, received at least 1 study vaccination, and provided immunogenicity data at Day 1 and Day 22, and who did not have any major protocol deviations that were assessed as potentially impacting on immunogenicity results.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- aQIV: MF59-adjuvanted Quadrivalent Subunit Inactivated Egg-derived Influenza Vaccine (aQIV) contains each of the 2 influenza type A strains and each of the 2 influenza type B strains in the vaccine.
Arm/Group | aQIV | aTIV-1 | aTIV-2
Number analyzed (Participants) | 872 | 436 | 433
Percentage of subjects
  A/H1N1 | 35.21 [32.03 to 38.48] | 39.45 [34.80 to 44.20] | 37.41 [32.8 to 40.20]
  A/H3N2 | 39.33 [36.08 to 42.67] | 39.70 [36.43 to 43.04] | 37.18 [32.6 to 41.9]
  B/Yamagata | 16.40 [14.0 to 19.03] | NA [NA to NA] — Not applicable as the strain is not present in an aTIV vaccine | 15.47 [12.2 to 19.2]
  B/Victoria | 13.42 [11.22 to 15.86] | 12.16 [9.24 to 15.60] | NA [NA to NA] — Not applicable as the strain is not present in an aTIV vaccine

4. Primary Outcome: Immunogenicity Endpoint: The Percent of Subjects Achieving an HI Antibody Titer ≥ 1:40 for the Four Strains Included in the Vaccines.
Description: The percentage of subjects vaccinated with aQIV achieving HI antibody titers ≥ 1:40 at Day 22 was assessed for each of the 4 strains. Assessment criteria was considered fulfilled if the lower bound of the two-sided 95% confidence interval for the percentage of subjects achieving a post-vaccination HI antibody titer ≥ 1:40 should meet or exceed 60%.
Time Frame: Day 22
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aQIV | aTIV-1 | aTIV-2
Number analyzed (Participants) | 872 | 436 | 433
Percentage of subjects
  A/H1N1 | 69.38 [66.20 to 72.43] | 71.79 [67.31 to 75.97] | 68.82 [64.23 to 73.16]
  A/H3N2 | 93.92 [92.12 to 95.41] | 94.72 [92.19 to 96.63] | 94.92 [92.41 to 96.79]
  B/Yamagata | 32.80 [29.69 to 36.03] | 21.79 [18.00 to 25.96] | 36.95 [32.39 to 41.69]
  B/Victoria | 38.19 [34.95 to 41.51] | 36.93 [32.38 to 41.65] | 24.48 [20.50 to 28.81]

5. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Titers (GMT) Against Homologous Strains
Description: For the assessment of GMTs using HI assay, aTIV-1 and aTIV-2 vaccine groups were pooled for the analysis of A-H1N1 and A-H3N2 strains. aTIV-1 and aTIV-2 vaccine groups are pooled for the analysis of A-H1N1 and A-H3N2 strains. For B-Victoria TIV=aTIV-1. For B-Yamagata TIV=aTIV-2.
  The immunologic superiority in HI antibody responses for the alternate B strain (eg, the influenza B strain included in the aQIV but not in the aTIV formulation) were assessed for each aTIV separately, using the GMT ratio (aTIV/aQIV) at Day 22.
Time Frame: Day 1 and Day 22
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | aQIV | aTIV-1 | aTIV-2 | aTIV-1/aTIV-2
Number analyzed (Participants) | 872 | 436 | 433 | 869
geometric mean titer
  A/H1N1 Day 1 | 19.07 [17.66 to 20.60] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 18.77 [17.47 to 20.17]
  A/H1N1 Day 22 | 57.07 [52.67 to 61.84] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 63.73 [58.60 to 69.32]
  A/H3N2 Day 1 | 73.27 [66.36 to 80.90] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 71.83 [65.39 to 78.90]
  A/H3N2 Day 22 | 245.85 [225.57 to 267.95] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 236.27 [217.53 to 256.63]
  B/Yamagata Day 1 | 10.41 [9.86 to 10.98] | NA [NA to NA] — Analysis not specified for alternate strain. | 10.76 [9.97 to 11.61] | NA [NA to NA] — Analysis was not performed.
  B/Yamagata Day 22 | 21.15 [19.75 to 22.66] | NA [NA to NA] — Analysis not specified for alternate strain. | 20.74 [18.86 to 22.80] | NA [NA to NA] — Analysis was not performed.
  B/Victoria Day 1 | 14.15 [13.30 to 15.05] | 15.18 [13.85 to 16.64] | NA [NA to NA] — Analysis not specified for alternate strain. | NA [NA to NA] — Analysis was not performed.
  B/Victoria Day 22 | 24.91 [23.21 to 26.74] | 25.54 [23.03 to 28.33] | NA [NA to NA] — Analysis not specified for alternate strain. | NA [NA to NA] — Analysis was not performed.
Statistical Analysis 1: Comparison: aQIV vs aTIV-1; B/Yamagata strain: GMT Ratio (aTIV/aQIV); Test type: Superiority — Superiority of aQIV vs. aTIV-1 for the alternate B strain was assessed using the GMT ratio (GMTaTIV/GMTaQIV); Superiority was declared if the upper limit of the two-sided 95% CI for the GMT ratio (aTIV/aQIV) was <1. The superiority comparison was based on the Full Analysis Set (FAS) Immunogenicity comprised all subjects who were randomized, received at least 1 study vaccination, and provided immunogenicity data at Day 1 and Day 22; GMT ratio = 0.64, 95% CI 2-sided [0.58 to 0.70]
Statistical Analysis 2: Comparison: aQIV vs aTIV-2; B/Victoria Strain: GMT Ratio (aTIV/aQIV); Test type: Superiority — Superiority of aQIV vs. aTIV-2 for the alternate B strain was assessed using the GMT ratio (GMTaTIV/GMTaQIV); Superiority was declared if the upper limit of the two-sided 95% CI for the GMT ratio (aTIV/aQIV) was <1. The superiority comparison was based on the FAS Immunogenicity; GMT ratio = 0.71, 95% CI 2-sided [0.64 to 0.78]

6. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) of Post Vaccination HI Titer Over the Pre-vaccination HI Titer Against Homologous Strains
Description: The GMR was assessed as the postvaccination HI titer divided by the prevaccination HI titer (Day 22/Day 1). aTIV-1 and aTIV-2 vaccine groups were pooled for the analysis of A-H1N1 and A-H3N2 strains. For B-Victoria TIV=aTIV-1. For B-Yamagata TIV=aTIV-2.
Time Frame: Day 22/Day 1
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean ratio
Arm/Group | aQIV | aTIV-1 | aTIV-2 | aTIV-1/aTIV-2
Number analyzed (Participants) | 872 | 436 | 433 | 869
geometric mean ratio
  A/H1N1 | 2.99 [2.78 to 3.22] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 3.40 [3.14 to 3.67]
  A/H3N2 | 3.36 [3.07 to 3.66] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 3.29 [3.02 to 3.59]
  B/Yamagata | 2.03 [1.92 to 2.15] | NA [NA to NA] — Analysis not specified for alternate strain. | 1.93 [1.79 to 2.08] | NA [NA to NA] — Analysis was not performed.
  B/Victoria | 1.76 [1.66 to 1.86] | 1.68 [1.55 to 1.82] | NA [NA to NA] — Analysis not specified for alternate strain. | NA [NA to NA] — Analysis was not performed.

7. Secondary Outcome: Immunogenicity Endpoint: The Percentage of Subjects With a Titer ≥1:40 Against Homologous Strains
Description: The percentage of subjects with HI titer of ≥1:40 at Day 1 (prevaccination) and Day 22 (postvaccination) was assessed for homologous strains. aTIV-1 and aTIV-2 vaccine groups are pooled for the analysis of A-H1N1 and A-H3N2 strains. For B/Victoria TIV=TIV-1. For B/Yamagata TIV=TIV-2.
Time Frame: Day 1 and Day 22
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV | aTIV-1 | aTIV-2 | aTIV-1/aTIV-2
Number analyzed (Participants) | 872 | 436 | 433 | 869
percentage of subjects
  A/H1N1 Day 1 | 33.26 [30.13 to 36.49] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 31.07 [28.00 to 34.27]
  A/H1N1 Day 22 | 69.38 [66.20 to 72.43] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 70.31 [67.15 to 73.33]
  A/H3N2 Day 1 | 70.64 [67.50 to 73.65] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 70.66 [67.50 to 73.67]
  A/H3N2 Day 22 | 93.92 [92.12 to 95.41] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 94.82 [93.13 to 96.20]
  B/Yamagata Day 1 | 11.12 [9.11 to 13.40] | NA [NA to NA] — Analysis not specified for alternate strain. | 11.55 [8.69 to 14.94] | NA [NA to NA] — Analysis was not performed.
  B/Yamagata Day 22 | 32.80 [26.69 to 36.03] | NA [NA to NA] — Analysis not specified for alternate strain. | 36.95 [32.39 to 41.69] | NA [NA to NA] — Analysis was not performed.
  B/Victoria Day 1 | 19.72 [17.13 to 22.52] | 22.71 [18.86 to 26.93] | NA [NA to NA] — Analysis not specified for alternate strain. | NA [NA to NA] — Analysis was not performed.
  B/Victoria Day 22 | 38.19 [34.95 to 41.51] | 36.93 [32.38 to 41.65] | NA [NA to NA] — Analysis not specified for alternate strain. | NA [NA to NA] — Analysis was not performed.

8. Secondary Outcome: Immunogenicity Endpoint: The Percentage of Subjects With SCR Against Homologous Strains
Description: The SCR was defined as the percentage of subjects with either a prevaccination HI titer <1:10 and a postvaccination HI titer ≥1:40 or a prevaccination HI titer ≥1:10 and a ≥4-fold increase in postvaccination HI titer. For assessment if SCR using HI assay, aTIV-1 and aTIV-2 vaccine groups were pooled for the analysis of A-H1N1 and A-H3N2 strains. For B-Victoria TIV=aTIV-1. For B-Yamagata TIV=aTIV-2.
  The immunologic superiority in HI antibody responses for the alternate B strain (eg, the influenza B strain included in the aQIV but not in the aTIV formulation) were assessed for each aTIV separately, using the difference in SCR (aTIV-aQIV) at Day 22.
Time Frame: Day 22
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aQIV | aTIV-1 | aTIV-2 | aTIV-1/aTIV-2
Number analyzed (Participants) | 872 | 436 | 433 | 869
Percentage of subjects
  A/H1N1 | 35.21 [32.03 to 38.48] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 38.43 [35.19 to 41.76]
  A/H3N2 | 39.33 [36.08 to 42.67] | NA [NA to NA] — Analysis not specified for individual strain. | NA [NA to NA] — Analysis not specified for individual strain. | 39.70 [36.43 to 43.04]
  B/Yamagata | 16.40 [14.00 to 19.03] | NA [NA to NA] — Analysis not specified for alternate strain. | 15.47 [12.20 to 19.23] | NA [NA to NA] — Analysis was not performed.
  B/Victoria | 13.42 [11.22 to 15.86] | 12.16 [9.24 to 15.60] | NA [NA to NA] — Analysis not specified for alternate strain. | NA [NA to NA] — Analysis was not performed.
Statistical Analysis 1: Comparison: aQIV vs aTIV-1; B/Yamagata Strain: SCR Difference (aTIV-1 - aQIV); Test type: Superiority — Superiority of aQIV vs. aTIV-1 for the alternate B strain was assessed using the difference in SCR (SCRaTIV-SCRaQIV) at Day 22. Superiority was declared if the upper limit of the two-sided 95% CI for the difference in SCRs (aTIV-aQIV) was <0, for both B strains. The superiority comparison was based on the FAS Immunogenicity; SCR difference = -11.96, 95% CI 2-sided [-15.12 to -8.81]
Statistical Analysis 2: Comparison: aQIV vs aTIV-2; B/Victoria Strain: SCR Difference (aTIV-2 - aQIV); Test type: Superiority — Superiority of aQIV vs. aTIV-2 for the alternate B strain was assessed using the difference in SCR (SCRaTIV-SCRaQIV) at Day 22. Superiority was declared if the upper limit of the two-sided 95% CI for the difference in SCRs (aTIV-aQIV) was <0, for both B strains. The superiority comparison was based on the FAS Immunogenicity; SCR difference = -10.82, 95% CI 2-sided [-13.54 to -8.11]

9. Secondary Outcome: Safety Endpoint: Number of Subjects With Solicited Local and Systemic Adverse Events (AEs) Following Vaccination
Description: Safety of vaccination was assessed in terms of percentage of subjects reporting solicited AEs up to 7 days after vaccination.
Time Frame: Day 1 through Day 7
Population: The Solicited Safety Set consists of all subjects in the FAS who received at least one dose or partial dose of study vaccine and have provided any evaluable follow-up safety data (solicited AE data).
Measure: Count of Participants; unit: Participants
Arm/Group | aQIV | aTIV-1 | aTIV-2
Number analyzed (Participants) | 883 | 439 | 438
Participants
  Any local solicited AE | 385 | 170 | 167
  Any systemic solicited AE | 231 | 107 | 110

10. Secondary Outcome: Safety Endpoint: Number of Subjects With Unsolicited AEs
Description: Safety of vaccination was assessed in terms of percentage of subjects reporting unsolicited AEs up to 21 days after vaccination.
Time Frame: Day 1 through Day 22
Population: The Overall Safety Set consists of all subjects in the FAS who received at least one dose or partial dose of study vaccine and have provided any evaluable follow-up safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | aQIV | aTIV-1 | aTIV-2
Number analyzed (Participants) | 888 | 444 | 444
Participants | 136 | 50 | 68

11. Secondary Outcome: Safety Endpoint: Number of Subjects With Serious AEs (SAEs), AEs Leading to Withdrawal From the Study, New Onset of Chronic Diseases (NOCDs) and AEs of Special Interest (AESIs)
Description: Safety of vaccination was assessed in terms of percentage of subjects reporting SAEs, AEs leading to withdrawal, NOCDs, and AESIs and medically attended AE up to 180 days after vaccination.
Time Frame: Day 1 through Day 181
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | aQIV | aTIV-1 | aTIV-2
Number analyzed (Participants) | 888 | 444 | 444
Participants
  SAEs | 37 | 28 | 18
  AEs leading to withdrawal | 0 | 0 | 0
  NOCDs | 23 | 16 | 14
  AESIs | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: SAEs and unsolicited AEs: Day 1 through 181; Solicited AEs: Day 1 through 7
Arm/Group | aQIV | aTIV-1 | aTIV-2
All-Cause Mortality (participants affected / at risk) | 2/888 | 0/444 | 0/444
Serious Adverse Events (participants affected / at risk) | 37/888 | 28/444 | 18/444
Other Adverse Events (participants affected / at risk) | 461/888 | 217/444 | 215/444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV (N=888) | aTIV-1 (N=444) | aTIV-2 (N=444)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 7 | 4 | 1
Influenza (Infections and infestations) | 1 | 0 | 2
Sepsis (Infections and infestations) | 1 | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Viral pericarditis (Infections and infestations) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 2 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV (N=888) | aTIV-1 (N=444) | aTIV-2 (N=444)
Redness (General disorders) | 188 | 77 | 81
Swelling (General disorders) | 134 | 69 | 64
Pain (General disorders) | 275 | 125 | 109
Fatigue (General disorders) | 144 | 67 | 52
Myalgia (Musculoskeletal and connective tissue disorders) | 71 | 34 | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 80 | 37 | 31
Headache (Nervous system disorders) | 105 | 46 | 49
Diarrhea (Gastrointestinal disorders) | 48 | 24 | 30
Ecchymosis (General disorders) | 69 | 28 | 23
Other (General disorders) | 48 | 12 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT03314662/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03314662/SAP_001.pdf